CLINICAL TRIAL: NCT05256693
Title: Prevention of C.Difficile Infections With Oral Vancomycine in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant: a Double-blind Placebo-controlled Randomized Clinical Trial
Brief Title: Prevention of C.Difficile Infections With Oral Vancomycine in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplant
Acronym: VANCALLO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GIRCI Ile de France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APHP210089
Record Dates: First submitted 2022-01-28; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-11

CONDITIONS: Clostridium Difficile Infections; Stem Cell Transplant Complications
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vancomycine (Experimental): Oral vancomycine 125 mg twice a day, from inclusion (at the time of hospitalization for allogeneic stem cell transplant) until hospital discharge or 5 weeks in hospital at most.
  Interventions: Drug: Vancomycin
- Placebo (Placebo Comparator): Vancomycine placebo, twice a day, from inclusion (at the time of hospitalization for allogeneic stem cell transplant) until hospital discharge or 5 weeks in hospital at most.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin — Oral vancomycin (powder) 125mg twice a day
  Arms: Vancomycine
Drug: Placebo — Vancomycine placebo (powder) twice a day
  Arms: Placebo

SUMMARY:
Clostridium difficile (CD) infection are an important cause of morbi-mortality in patients undergoing allogeneic hematopoietic stem cell transplant (HSCT). The VANCALLO trial aims at evaluating oral vancomycine reducing the risk of CD infection relying on a placebo controlled 1:1 randomized design, including one interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥15 ans
* Hospitalization since less than 72 hours, for an allogeneic stem cell transplant, whichever the indication and conditioning
* For men and women of reproductive age: use of contraceptives
* Informed consent
* Healthcare insurance

Exclusion Criteria:

* Know allergy or history of adverse events with vancomycine
* Pregnancy
* Clostridium difficile infection within 30 days prior to inclusion or at inclusion
* History of total colectomy and/or inflammatory bowel disease
* Progressive diarrhea at inclusion, whichever the etiology
* Digestive decontamination protocol for the stem cell transplant procedure
* Participation to another drug clinical trial or being in the exclusion period from a prior clinical trial participation

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Clostridium difficile infection | 5 weeks
  Clostridium difficile infection defined as a diarrhea (> 3 loose stools/day) with positive Clostridium difficile testing and free-toxin in stools by enzyme-linked immunosorbent assay (ELISA), without other obvious etiology for diarrhea nor pseudo-membraneous colitis (endoscopy, colectomy, autopsy).

SECONDARY OUTCOMES:
Proportion of patients with Clostridium difficile infection | 12 weeks
  Clostridium difficile infection defined as a diarrhea (> 3 loose stools/day) with positive Clostridium difficile testing and free-toxin in stools by enzyme-linked immunosorbent assay (ELISA), without other obvious etiology for diarrhea nor pseudo-membraneous colitis (endoscopy, colectomy, autopsy).
Cumulative incidence of Clostridium difficile infection | 5 weeks
  Time between inclusion and Clostridium difficile infection, occurring before hospital discharge or the end of study treatment (that is 5 weeks from inclusion if the patient is still hospitalized), defined as a diarrhea (> 3 loose stools/day) with positive Clostridium difficile testing and free-toxin in stools by enzyme-linked immunosorbent assay (ELISA), without other obvious etiology for diarrhea nor pseudo-membraneous colitis (endoscopy, colectomy, autopsy).
Proportion of patients with Clostridium difficile infection by PCR testing | 5 weeks
  Clostridium difficile infection defined as a diarrhea (> 3 loose stools/day) with positive toxinogenic Clostridium difficile PCR (polymerase chain reaction) testing, without other obvious etiology for diarrhea nor pseudo-membraneous colitis (endoscopy, colectomy, autopsy).
Factors associated with the proportion of patients with Clostridium difficile infection | 5 weeks
  Candidate factors associated with Clostridium difficile infection: antibiotics, toxinogenic strain at baseline, microbiota composition
Proportion of patients with severe Clostridium difficile infection | 5 weeks
  Severe Clostridium difficile infection defined as at least one of the following: fulminans colitis, toxic megacolon, dehydration, neutrophils blood count>20000/mm3, general deterioration
Proportion of patients with bacterial infection | 5 weeks
  Bacterial infection defined as occurrence of a bacterial infection (any site)
Proportion of patients with vancomycin-resistant enterococcus carriage | 5 weeks
  Carriage defined as occurrence of vancomycin-resistant enterococcus carriage on rectal swab
Gut microbiome profile | 12 weeks
  Evolution of gut microbiome profile during the study
Nosocomial Clostridium difficile infection clusters | 12 weeks
  Defined as at least 2 cases of Clostridium difficile infection in the department within 12 weeks
Proportion of patients with Graft-versus-Host disease | 12 months
  Graft-versus-Host disease, acute or chronic, grade 2 to 4
Cumulative incidence of relapse | 12 months
  Time between inclusion and hemopathy relapse or last follow-up, up to a maximum of 12 months
Treatment-related mortality | 5 weeks
  Proportion of death related to allogeneic stem cell transplant procedures
Overall survival | 12 months
  Time between inclusion and death or last follow-up, up to a maximum of 12 months

IPD SHARING:
Plan to Share IPD: Undecided